CLINICAL TRIAL: NCT03350152
Title: Treatment With Low-Dose Cytarabine in Elderly Patients (Age 70 Years or Older) With Acute Myeloid Leukemia: A Single Institution Experience.
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: HCL
Record Dates: First submitted 2017-11-08; First posted 2017-11-22 (Actual); Last update posted 2017-11-22 (Actual); Status verified 2017-10

CONDITIONS: Acute Myeloid Leukemia
Keywords: Chemotherapy, Low-intensity therapy, elderly, prognosis,
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LAM group: Have a diagnosis of AML according to World Health Organization (WHO) classification Are at least 70 years of age

SUMMARY:
The treatment of very elderly patients (≥70 years) with acute myeloid leukemia remains controversial. Although the outcome in younger adults has improved because of cytarabine- and anthracycline-based chemotherapy with advanced supportive care and introduction of hematopoietic stem cell transplantation, the benefit associated with standard intensive chemotherapy in older patients remain debatable. Life expectancy in elderly patients is a function of age, disability and comorbidity, performance score, along with leukemia characteristics such as genetic alterations or white blood cell count at diagnosis 'Older' patients are generally considered those aged 60 years or older.

Intensive chemotherapy delivered to the very elderly with AML (patients _70 years of age), may not be beneficial to most and could be harmful to some. However, these patients are often referred to as 'unfit' or ineligible for intensive remission induction therapy. In daily practice, the final decision to treat intensively or not is made by the treating hematologist on a case by case basis according to patient's age, cytogenetics, performance score, concomitant diseases and type of AML (de novo or secondary).

In older patients considered 'unfit' for intensive treatment, LD-AraC has been demonstrated to be more beneficial than best supportive care and hydroxyurea. The recent availability of new drugs that may have an improved side effect profile and in some cases bioavailability may offer future improvement for this patient population. The efficacy of hypomethylating agents has been studied in older AML patients with conflicting results. Recent publications refined prognostic information, which not only optimize existing treatments but also could lead to the development of additional targeted therapeutic approaches.

In this study, the investigators focus on patients with AML (_20% blasts) aged 70 or older seen in our institution over a 14-year period. The objectives of the analysis are to describe the demographic, clinical and biological characteristics of this population and to evaluate how these characteristics and the treatment chosen affect

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of AML according to World Health Organization (WHO) classification
* Are at least 70 years of age

Exclusion Criteria:

- Patients with M3 AML of FAB classification (APL, Acute Promyelocytic Leukemia)

Age Groups: Child, Adult, Older Adult
Study Population: * Have a diagnosis of AML according to World Health Organization (WHO) classification
  * Are at least 70 years of age
  * Gender male and female
Sampling Method: Non-Probability Sample
Enrollment: 302 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2014-06-01 (Actual); Study Completion 2014-06-01 (Actual)

PRIMARY OUTCOMES:
overall survival (OS) | Date of last contact if alive, up to 100 months
  OS was the main endpoint for this analysis. The event for OS was death, and patients were censored at the date of last contact, if alive.

CONTACTS AND LOCATIONS:
Locations (1):
- CORTIAL, Pierre-Bénite, Rhone, France

IPD SHARING:
Plan to Share IPD: No